CLINICAL TRIAL: NCT00968929
Title: Efficacy and Safety Evaluation of Recombinant Streptokinase and Urokinase in the Treatment of Pulmonary Embolism: A Multi-Center, Randomized Controlled Trial in China
Brief Title: Recombinant Streptokinase Versus Urokinase in Pulmonary Embolism in China (RESUPEC)
Acronym: RESUPEC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Qingdao University (Other); Tianjin Medical University General Hospital (Other); General Hospital of Shenyang Military Region (Other); Guangdong Institute of Respiratory Disease (Unknown); The First Affiliated Hospital of Shanxi Medical University (Other); Shenzhen People's Hospital (Other); Ningxia Medical University (Other)
Responsible Party: Chen WANG, Beijing Institute of Respiratory Medicine, Beijing Chao-Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006BAI01A06
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Pulmonary Embolism; Pulmonary Thromboembolism
Keywords: pulmonary embolism; thrombolysis; massive; submassive; recombinant streptokinase; urokinase
MeSH Terms: conditions — Pulmonary Embolism | interventions — Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- r-SK group (Experimental): Recombinant streptokinase: 1.5 million IU continuously intravenous infusion for 2 hours
  Interventions: Drug: Recombinant Streptokinase
- UK group (Active Comparator): Urokinase: 20,000 IU/kg continuously intravenous infusion for 2 hours
  Interventions: Drug: Urokinase

INTERVENTIONS:
Drug: Recombinant Streptokinase — Recombinant streptokinase: 1.5 million IU continuously intravenous infusion for 2 hours
  Arms: r-SK group
Drug: Urokinase — Urokinase: 20,000 IU/kg continuously intravenous infusion for 2 hours
  Arms: UK group

SUMMARY:
Recombinant streptokinase (r-SK) is an effective thrombolytic agent developed with gene engineering. Its characteristics of high output and low production cost make it affordable in treating acute myocardial infarction (AMI) in developing countries. It is unclear whether r-SK can be used in patients with pulmonary embolism (PE). The aim of this study was to investigate the efficacy and safety of 1.5 million IU r-SK by 2 hours infusion and 20,000 IU/kg urokinase (UK) by 2 hours infusion in selected PE patients.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is a common cardiovascular illness. Massive PE is characterized with cardiogenic shock and/or persistent arterial hypotension. Submassive PE patients are defined with right ventricular dysfunction (RVD) identified by echocardiography or CT and the etc. The mortality of massive and submassive PE is higher than low-risk PE. PE has the mortality rate of >15% in the first 3 months after diagnosis. Thrombolytic treatment should be commenced as soon as possible after high-risk PE was diagnosed. Thrombolysis has been proved to be the most rapid and effective therapy to reduce the obstruction of pulmonary circulation and normalize hemodynamic parameters. The ultimate goals of thrombolytic therapy for this disease are to minimize early morbidity and mortality and to prevent recurrence without provoking excessive bleeding.

Currently, the choice of thrombolytic agents and regimens (SK, UK or rt-PA) is mostly based on personal or regional preferences. A novel dosing regimen of UK (3 million IU/2h, or 4400 IU/kg as a loading dose followed by 4400 IU/kg/h over 12h) and SK (1.5 million IU /2h) have been recommended in ESC guidelines. Considering lower body weight in Chinese population, a relative lower dosage UK-2h (20,000 IU/kg) regimen combined with low molecular weight heparin (LMWH) has been used in Chinese population. Our previous study has revealed that the efficacy and safety of UK-2h (20 000 IU/Kg) were similar with UK-12h (standard regimen) in Chinese patients. Thus the UK-2h (20,000 IU/Kg) became a popular and alternative choice in treating PE in China for its lower cost and convenience. Natural streptokinase (n-SK or SK) is an old thrombolytic agent. However, its immunogenicity lowers its safety and that constitute a concern among doctors. In recent years, as the development of gene engineering, r-SK was produced. R-SK has the advantage of not containing streptolysin and streptodornase unlike streptococci-derived n-SK which might make it safer theoretically. For its low cost, r-SK has been used to treat AMI especially in developing countries. In this study, the efficacy and safety between r-SK (1.5 million IU/2h) and UK-2h (20 000U/Kg) for treating acute PE will be compared. The study is conducted in patients with massive PE and submassive PE. The clinical efficacy, emboli dissolving efficacy and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic PTE confirmed either by CTPA or by a high probability ventilation-perfusion lung scanning (V/Q scan).
* Presented with hemodynamic instability (systolic blood pressure <90 mmHg or a fall in systolic blood pressure of more than 40 mmHg for at least 15 min, or cardiogenic shock) or associated with RVD identified by echocardiography or CT.
* Symptoms deterioration less than 14 days before diagnosis.

Exclusion Criteria:

* Active bleeding or spontaneous intracranial hemorrhage in the preceding 6 months
* Major surgery, organ biopsy or recent puncture of a non-compressible vessel in the preceding 2 weeks
* Cerebral arterial thrombosis in the preceding 2 months
* Gastro-intestinal bleeding in the preceding 10 days
* Major trauma within the past 15 days
* Neurosurgery or ophthalmologic operation in the preceding 1 month
* Uncontrolled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg)
* Recent external cardiac resuscitation manoeuvres
* Platelet count < 100,000/mm3 at admission
* Pregnancy, puerperium or lactation in the preceding 2 weeks
* Infectious pericarditis or endocarditis
* Severe hepatic and kidney dysfunction
* Hemorrhagic retinopathy due to diabetes
* A known bleeding disorder.
* Chronic thromboembolic pulmonary hypertension (CTEPH) without new pulmonary thromboembolism (PTE)
* Received streptokinase in the preceding 6 months
* Infected by streptococcus in the preceding 1 month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2006-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The improvement of the right ventricular function on echocardiogram | within the 1st, 14 days and 3 months
Quantitative computed tomographic pulmonary angiography (CTPA) score | 1st, 14 days and 3 months
The relief of symptoms | 2-4h, 1st, 4th , 7th, 10th, 14 days day and 3 months

SECONDARY OUTCOMES:
Major or minor bleeding | 14 days and 3 months
Pulmonary embolism recurrence | 14 days and 3 months
Death | 14 days and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Chen WANG, Prof, Principal Investigator — Beijing Institute of Respiratory Medicine, Beijing-Chao Yang Hospital
Locations (8):
- China (8):
  - Beijing Institute of Respiratory Medicine, Beijing Chao-Yang hospital, Beijing, Beijing Municipality
  - Guangdong Institute of Respiratory Disease, Guangzhou Medical University,, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The General Hospital of Shenyang Military Command, Shenyang, Liaoning
  - Affiliated Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao, Shandong
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Background] Zhu L, Yang Y, Wu Y, Zhai Z, Wang C. Value of right ventricular dysfunction for prognosis in pulmonary embolism. Int J Cardiol. 2008 Jun 23;127(1):40-5. doi: 10.1016/j.ijcard.2007.06.093. Epub 2007 Aug 22. PMID 17716753
- [Background] Zhu L, Yang YH, Wu YF, Zhai ZG, Wang C; National Project of the Diagnosis and Treatment Strategies for Pulmonary Thromboembolism investigators. Value of transthoracic echocardiography combined with cardiac troponin I in risk stratification in acute pulmonary thromboembolism. Chin Med J (Engl). 2007 Jan 5;120(1):17-21. PMID 17254482
- [Background] Zhu L, Wang C, Yang Y, Wu Y, Zhai Z, Dai H, Pang B, Tong Z. Value of transthoracic echocardiography in therapy regimens evaluation in pulmonary embolism. J Thromb Thrombolysis. 2008 Dec;26(3):251-6. doi: 10.1007/s11239-007-0087-8. Epub 2007 Aug 21. PMID 17705052
- [Background] Yang Wang, Chen Wang, Yuanhua Yang, Baosen Pang. Effect of recombinant single-chain urokinase-type plasminogen activator on experimental pulmonary embolism. Clin Appl Thromb Hemost. 2010 Oct;16(5):537-42. doi: 10.1177/1076029609343003. Epub 2009 Oct 14. PMID 19833628